CLINICAL TRIAL: NCT05881954
Title: Early Outcomes of Natives and Graft-related Femoral Reconstruction Managed With Orthotopic Xenopericardial Patchs
Brief Title: Outcomes of Natives and Graft-related Femoral Reconstruction With Tubulized Pericardial Patchs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Hostalrich Aurelien, MD, Clinical Professor, University Paul Sabatier of Toulouse
Other Study IDs: FEMORALROLLED
Record Dates: First submitted 2023-04-28; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Vascular Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Groin infection — Femoral artery reconstruction with tubulized pericardium patch

SUMMARY:
Groin wound infection after arterial femoral prosthetic reconstruction or percutaneous access and drug abusers are frequent and increase largely the post operative morbi-mortality.

There is no perfect substitute to replace infected graft or to restaure femoral artery in septic condition moreover when all the femoral bifurcation is involved with a femoro-femoral bypass mandatory.

Seeing the encouraging results of rolled pericardium patch to treat native and prosthetics aortic infections in term of patency and infection resistance, the investigators propose to evaluate the outcomes of this subsitute rolled with samples in case of femoro-femoral repair in septic condition.

DETAILED DESCRIPTION:
Groin wound infection after vascular surgery is a frequent complication with a significant increase in post operative morbidity and mortality. Actual studies reported more than 20% of patients who develop groin wound infection with an important rate of reintervention and risk in limb loss. Theses groin complications are frequent in drug abusers but can also happen after percutaneous femoral access for endovascular therapy leading to arterial reconstruction.

After mechanical debridement and eventually muscle flap rotation, ESVS 2020 guidelines recommend in situ reconstruction with the use of autogenous reconstruction vein femoral vein but it is a demanding surgery especially in redo surgery with extensive incision and deep venous complication. Saphenous vein is often too small in diameter to perform a femoro-femoral reconstruction. The other possibility is cryopreserved Cadaveric Arterial Allograft which are difficult to obtain in sufficient time for an urgent operation with frequent aneurysmal evolution. Literature reports up to 30% of reinfection with rifampin-soaked Dacron conduit are used with frequent reintervention. Rolled Bovine pericardium grafts have been proposed as a primary intention substitute in native and prosthetics aortic infections and are presented as resistant to infection when used as patch repair in case of groin complications. The aim of our study was to evaluate the outcomes in term of patency, limb salvage and infection resistance of this substitute when tubulized with stample in groin wound infection to replace previous prosthetic graft with active infection or false aneurysm rupture or after percutaneous septic femoral access complication in emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* Previous femoral artery reconstruction with infected graft
* Femoral artery septic false aneurysm needed complete arterial reconstruction (drug abuser or percutaneous femoral access)

Exclusion Criteria:

* Simple patch closure of femoral artery
* Groin infection without femoral artery reconstruction Pregnancy Minors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting a graft infection in the groin or a septic false aneurysm of the femoral artery.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Patency | 3 months
  Patency of the bypass
Absence of reinfection | After antibiotherapy (6 weeks generally)
  Disparition of infections signs : biological and clinically

SECONDARY OUTCOMES:
Reintervention | 30 days post operative; 3 months, 6 months, 12 months
  Need of reoperation during the follow up
Late patency | 6 months
  Patency of the Bypass

CONTACTS AND LOCATIONS:
Locations (1):
- Aurélien Hostalrich [ahostalrich], Toulouse, France

REFERENCES:
- [Background] Alonso W, Ozdemir B, Chassin-Trubert L, Ziza V, Alric P, Canaud L. Early outcomes of native and graft-related abdominal aortic infection managed with orthotopic xenopericardial grafts. J Vasc Surg. 2021 Jan;73(1):222-231. doi: 10.1016/j.jvs.2020.04.513. Epub 2020 May 20. PMID 32442610
- [Background] McMillan WD, Leville CD, Hile CN. Bovine pericardial patch repair in infected fields. J Vasc Surg. 2012 Jun;55(6):1712-5. doi: 10.1016/j.jvs.2011.11.139. Epub 2012 Mar 28. PMID 22459752